CLINICAL TRIAL: NCT04864236
Title: A Randomized Controlled Trial to Test a Novel Negative Pressure Isolation Device During Aerosol Generating Procedures in the Operating Room
Brief Title: An Isolation Device to Contain Aerosol During Aerosol Generating Procedures in the Operating Room
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: John Shin (Other)
Responsible Party: Sponsor-Investigator, John Shin, Assistant Clinical Professor of Anesthesiology, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-000022
Record Dates: First submitted 2021-04-19; First posted 2021-04-28 (Actual); Results first posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-09

CONDITIONS: Aerosol Containment; Aerosol Generating Procedure
Keywords: health care worker exposure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Intervention group (Experimental): This group will undergo airway management in the operating room as part of the anesthesia for surgery in the presence of the novel isolation device.
  Interventions: Device: Novel isolation device to contain aerosol
- Control group (No Intervention)

INTERVENTIONS:
Device: Novel isolation device to contain aerosol — The novel isolation device is called SLACC (Suction-assisted Local Aerosol Containment Chamber). SLACC has the ability to isolate the atmosphere around the patient's upper airway (nose, mouth, throat) via negative pressure in a manner analogous to isolation rooms used to house patients with communicable diseases spread by aerosol (e.g. tuberculosis).
  The SLACC uses an external suction source to maintain a negative pressure micro-atmosphere around a patient's head (the source of infectious aerosols). The components of SLACC include a clear polymer frame, a flexible drape, and integrated sealed arm sleeves to protect the hands and forearms of the health care provider. The structure is flexible during use, transparent, can be rapidly assembled, and easily collapsible for removal and transport. Once deployed with the patient's head inside the chamber, the drape is secured across the open side of the chamber with adhesive and covers the patient's torso.
  Arms: Intervention group

SUMMARY:
The purpose of this study is to test the safety and efficacy of a new isolation device to contain aerosol during aerosol-generating procedures in the operating room.

DETAILED DESCRIPTION:
Patients with SARS-CoV-2 infections may require procedures that generate infectious aerosols (suspension of tiny particles or droplets in the air). Aerosols are believed to be the primary method of spread of SARS-CoV-2, as well as many other communicable diseases. In the health care setting, the providers who are in close proximity to patients during these aerosol-generating procedures (ie. Intubation (tube in your throat to help you breathe), noninvasive positive pressure ventilation (breathing support administered through a face or nasal mask) methods such as continuous positive airway pressure (CPAP) or bilevel positive airway pressure (BiPAP), bronchoscopy (thin tube through nose or mouth into the lungs), high flow nasal cannula (oxygen delivery through the nose at a very high flow rate)) are at risk for becoming infected with SARS-CoV-2. The current standard of care to prevent the spread of virus to health care workers involves the use of N-95 respirators (particulate filtering facepiece respirators), which have been intermittently in short supply throughout the current COVID-19 pandemic. In addition, even when there are adequate supplies of N-95 respirators, health care workers have been reusing the respirators multiple times, which may result in decreased efficacy and potential viral exposure. In order to provide enhanced protection to health care workers during aerosol-generating procedures, the study investigators have created a device, named SLACC (Suction-assisted Local Aerosol Containment Chamber). SLACC has the ability to isolate the atmosphere around the patient's upper airway (nose, mouth, throat) via negative pressure in a manner analogous to isolation rooms used to house patients with communicable diseases spread by aerosol (e.g. tuberculosis). Furthermore, SLACC is inexpensive, portable, and relatively simple to manufacture.

The SLACC uses an external suction source to maintain a negative pressure micro-atmosphere around a patient's head (the source of infectious aerosols). The components of SLACC include a clear polymer frame, a flexible drape, and integrated sealed arm sleeves to protect the hands and forearms of the health care provider. The structure is flexible during use, transparent, can be rapidly assembled, and easily collapsible for removal and transport. It is assembled using adhesive-backed polymer sections, allowing the structure to fold from a flat shipping/storage conformation into a free-standing structure. Once deployed with the patient's head inside the chamber, the drape is secured across the open side of the chamber with adhesive and covers the patient's torso. Many other containment devices have been proposed during the COVID-19 pandemic, but none have been demonstrated to contain aerosols effectively. With external suction applied, the investigators believe SLACC vastly improves upon the aerosol containment ability of other devices. The investigators have tested SLACC in a simulated setting and recently published the results in a high-quality, peer-reviewed journal (PMID: 32541251).

The investigators propose to test the safety and efficacy of SLACC in containing contamination during aerosol-generating procedures in the operating room through a randomized controlled trial. The investigators have identified a method of objectively quantifying health care worker exposure to respiratory particles and plan to compare exposure to the number and size of respiratory particles when SLACC is used compared to the current standard of care (no device used).

ELIGIBILITY:
Inclusion Criteria:

* Elective scheduled surgery (not emergent)
* Planned general anesthesia requiring intubation

Exclusion Criteria:

* Patients refusing or unable to consent for any reason, including claustrophobia or inability to cooperate
* Patients predicted to require the use of fiberoptic bronchoscopy for intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Shin, MD, Principal Investigator — University of California Los Angeles Department of Anesthesiology
Locations (1):
- UCLA Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seger CD, Wang L, Dong X, Tebon P, Kwon S, Liew EC, Marijic J, Umar S, Hoftman NN. A Novel Negative Pressure Isolation Device for Aerosol Transmissible COVID-19. Anesth Analg. 2020 Sep;131(3):664-668. doi: 10.1213/ANE.0000000000005052. PMID 32541251

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: This group will undergo airway management in the operating room as part of the anesthesia for surgery in the presence of the novel isolation device.
  Novel isolation device to contain aerosol: The novel isolation device is called SLACC (Suction-assisted Local Aerosol Containment Chamber). SLACC has the ability to isolate the atmosphere around the patient's upper airway (nose, mouth, throat) via negative pressure in a manner analogous to isolation rooms used to house patients with communicable diseases spread by aerosol (e.g. tuberculosis).
  The SLACC uses an external suction source to maintain a negative pressure micro-atmosphere around a patient's head (the source of infectious aerosols). The components of SLACC include a clear polymer frame, a flexible drape, and integrated sealed arm sleeves to protect the hands and forearms of the health care provider. The structure is flexible during use, transparent, can be rapidly assembled, and easily collapsible for removal and transport. Once deployed with the patient's head inside the chamber, the drape is secured across the open side of the chamber with adhesive and covers the patient's torso.
- Control Group: This group will undergo airway management in the same manner as described for the intervention group except that there is no SLACC device.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 39 | 40
Completed | 39 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control Group: This group will undergo airway management in the operating room in an identical manner to the intervention group except that the SLACC device will not be used.
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 39 | 40 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 22 | 53
  >=65 years | 8 | 18 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (16.0) | 54.1 (19.3) | 52.9 (17.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 43
  Male | 16 | 20 | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 39 | 40 | 79

OUTCOME MEASURES:

1. Primary Outcome: Particle Count Measurements During Intubation
Description: particle counts will be measured using a commercially-available particle counter at two locations: at the level of the anesthesiology provider's face (at the patient's head), and at the level of the assistant provider's face (at the patient's side)
Time Frame: particle counts will be measured continuously from the time of patient's entry into the operating room until the patient has been intubated for surgery, approximately 15 minutes total
Measure: Median (Inter-Quartile Range); unit: particles/cm^3
Groups:
- Control Group: This group will undergo airway management as described for the intervention group, except that SLACC device will not be used.
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 39 | 40
particles/cm^3
  Deep breathing/coughing phase, patient location | 4026 [1778 to 7616] | 411 [211 to 987]
  Deep breathing/coughing phase, physician location | 105 [37 to 232] | 392 [207 to 1259]
  Deep breathing/coughing phase, assistant location | 74 [18 to 211] | 185 [98 to 302]
  Intubation phase, patient location | 1560 [728 to 3093] | 490 [235 to 1394]
  Intubation phase, physician location | 48 [15 to 145] | 556 [297 to 1579]
  Intubation phase, assistant location | 27 [5 to 80] | 218 [158 to 436]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Equivalence — We compared particle number counts between intervention and control groups using the Wilcoxon test. Analyses were conducted using IBM SPSS V28 and p-values <0.05 were considered statistically significant; p < 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Time to Intubation
Description: defined as time from the first entry of laryngoscope into pt's oropharynx to the time of confirmed successful tracheal intubation
Time Frame: during intubation
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Control Group: This group will undergo airway management in the same manner as described for the intervention group, except that the SLACC device will not be used.
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 39 | 40
seconds | 51.6 (22.2) | 41.8 (25.7)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Equivalence — Patient characteristics were summarized between groups using mean (SD) and formally compared using the t-test; p = 0.073, t-test, 1 sided

3. Secondary Outcome: Total Number of Intubation Attempts
Description: total number of intubation attempts during airway management
Time Frame: during intubation
Measure: Mean (Standard Deviation); unit: number of attempts
Groups:
- Control Group: This group will undergo airway management as described for the intervention group, except that the SLACC device will not be used.
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 39 | 40
number of attempts | 1.05 (0.22) | 1.08 (0.27)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Equivalence — Patient characteristics and study variables were summarized between groups using mean (SD) and formally compared using the t-test; p = 0.670, t-test, 1 sided

4. Secondary Outcome: Pre-operative Airway Assessment (Mallampati Score)
Description: Mallampati score, can be given a score of 1-4 (whole numbers only), score of 4 indicates higher likelihood of difficult intubation and score of 1 indicates lower likelihood of difficult intubation
Time Frame: pre-operative assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 39 | 40
score on a scale | 1.74 (0.68) | 1.53 (0.72)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Equivalence — Patient characteristics were summarized between groups using mean (SD) and formally compared using the t-test; p = 0.167, t-test, 1 sided

5. Secondary Outcome: Laryngoscopy Grade View (Cormack-Lehane) Obtained During Intubation
Description: Cormack-Lehane grade assigned by anesthesiologist during intubation, grade can be 1-4, grade 1 correlates with a view of entirety of vocal cords while grade 4 correlates with no view at all of any part of the vocal cords
Time Frame: during intubation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 39 | 40
score on a scale | 1.21 (0.41) | 1.10 (0.30)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Equivalence — Patient characteristics were summarized between groups using mean (SD) and formally compared using the t-test; p = 0.198, t-test, 1 sided

6. Secondary Outcome: Pre-operative Airway Assessment (Thyromental Distance)
Description: thyromental distance is the distance measured between the chin and the thyroid cartilage (both landmarks are readily palpable on physical exam), this distance is typically measured in centimeters or as a measure of the number of finger breadths (as reported here). Finger breadths is defined as the number of finger widths that can fit within the defined distance.
Time Frame: pre-operative assessment
Measure: Mean (Standard Deviation); unit: finger breadths
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 39 | 40
finger breadths | 3.10 (0.38) | 3.18 (0.45)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Equivalence — Patient characteristics were summarized between groups using mean (SD) and formally compared using the t-test; p = 0.442, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the patient's participation in the trial, which ended approximately 4 minutes after intubation (when all data stopped being collected). The course of a typical patient's participation in the trial averaged approximately 15 min.
Description: Additional adverse event data collected included failure to intubate and failure to complete airway management in the intervention group for any reason (patient refusal, surgeon refusal, anesthesiologist's clinical judgment).
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/40
Other Adverse Events (participants affected / at risk) | 0/39 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/36/NCT04864236/Prot_SAP_001.pdf